CLINICAL TRIAL: NCT00470509
Title: Adalimumab in Severe and Acute Sciatica
Acronym: ASAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Stephane Genevay, Dr, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASAS
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Sciatica
MeSH Terms: conditions — Sciatica | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adalimumab (Experimental): adalimumab (2 subcutaneous 40 mg injections on day 0 and 7)
  Interventions: Drug: Adalimumab
- Placebo (Placebo Comparator): 2 placebo injections on day 0 and 7
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Adalimumab — 2 subcutaneous injections on day 0 and 7
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebos — 2 subcutaneous injections on day 0 and 7
  Other Names: placebo injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether adalimumab (a TNF-alpha inhibitor) is effective in the treatment of severe and acute sciatica.

DETAILED DESCRIPTION:
Sciatica and low back pain are common problems that lead to major costs in Western countries. The presence of herniated disc is generally considered as the leading cause of sciatica. However, recent findings indicate that the presence of this mechanism is not sufficient to explain all the clinical signs of radiculopathy and that inflammatory mechanisms contribute also to the pathophysiology of sciatica. Indeed, herniated discs contain large amounts of tumor necrosis factor (TNF-alpha) which can induce acute and chronic inflammation and pain. It has recently been demonstrated that TNF-alpha inhibitors (infliximab or etanercept) were able to prevent the occurrence of pain in an experimental model of sciatica. In addition, two independent preliminary studies have shown that patients treated with TNF-alpha inhibitors had better evolution than an historical control group. This study has been designed to verify the hypothesis that TNF-alpha has a major role in human sciatica and that anti-TNF-alpha agents are interesting therapeutic approaches in severe sciatica.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients older than 18
2. Episode of radicular pain in one lower limb for less than 12 weeks.
3. Medical evaluation requiring hospitalisation because of pain or functional handicap
4. Patients presenting a characteristic leg pain in the L3, L4, L5, or S1 territories plus at least one of the following: :

   * positive straight-leg-raising test with an elevation of less than 70°
   * positive femoral stretched
   * clear clinical sign of nerve root involvement

     * muscle strength deficiency or
     * sensory disturbances in clear cut dermatome or
     * lower limb reflex asymmetry.
5. Oswestry score greater than 50
6. If there is a past history of radicular pain involving the same nerve root, a 6 months interval free of leg pain is required.
7. A confirmed herniated disc on usual imaging techniques (CT scan or MRI) in the vicinity of the clinically involved nerve root that has been performed within the last 2 years.
8. Written informed consent

Exclusion Criteria:

1. The presence of recent (<48 hours) severe muscle weakness (<3/5) or clinical signs of cauda equina compression, requiring immediate surgery.

   * If surgical procedure is required but is denied, either because of surgeon's decision or because of patient's fully informed decision, then this patient could be included in the protocol.
2. Comorbidities such as :

   * Coexisting infections (Chest X-ray will be performed to all patients and tuberculin skin test in case of doubt concerning a past history of tuberculous infection).
   * Autoimmune disease (other than RA).
   * History of cancer or malign lymphoproliferative disorders (unless the patient has been declared in remission for more than 5 years)
   * History of demyelinating disorders.
3. Pregnancy.
4. History of intolerance to adalimumab or any of its ingredients
5. Previous participation in this clinical study.
6. Participation in another clinical study within 4 weeks prior to the start of or during this study.
7. Poor motivation or other emotional or intellectual problems that are likely to limit the ability of the patient to comply with the protocol requirements.
8. The use of cortisone prior to the inclusion IS NOT an exclusion criteria

The investigators will also be allowed to exclude an individual patient from the study and remove the blinding in case of a superimposed infection or any severe side effect during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2005-05; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Leg pain | 6 months
  Evolution of leg pain over time. Pain will be assessed using a Visual Analog Scale (VAS).

SECONDARY OUTCOMES:
delta VAS | 6 months
  Percentage of amelioration for VAS and ODI (Oswestry Disability Index)
SF-12 | 6 months
  Assessment of patient's statisfaction and expectations using the SF12 general health questionnaire.
delta ODI | 6 months
  Percentage of amelioration for ODI (Oswestry Disability Index)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Genevay, MD, Principal Investigator — Geneva University Hospital & Swiss Society of Rheumatology
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Derived] Genevay S, Viatte S, Finckh A, Zufferey P, Balague F, Gabay C. Adalimumab in severe and acute sciatica: a multicenter, randomized, double-blind, placebo-controlled trial. Arthritis Rheum. 2010 Aug;62(8):2339-46. doi: 10.1002/art.27499. PMID 20506391